CLINICAL TRIAL: NCT03441204
Title: REgistry-based Randomized Controlled Trial of Treatment Duration and Mortality in Long-term OXygen Therapy (REDOX) A Multicenter, Phase IV, Registry-Based, Randomized Controlled Trial (R-RCT)
Brief Title: REgistry-based Treatment Duration and Mortality in Long-term OXygen Therapy (REDOX)
Acronym: REDOX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Skane University Hospital (Other)
Collaborators: Lund University (Other); Blekinge County Council Hospital (Other)
Responsible Party: Principal Investigator, Magnus Ekström, Principal Investigator, Skane University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REDOX 2016
Record Dates: First submitted 2018-02-01; First posted 2018-02-22 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Chronic Respiratory Failure With Hypoxia
Keywords: COPD; Long-term oxygen therapy (LTOT); Registry; Registry-based randomized controlled trial (R-RCT); Treatment duration; Mortality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTOT 24 h/day (intervention) (Active Comparator): Long-term oxygen therapy (LTOT) prescribed 24 h/day. The LTOT is provided according to standard clinical practice using oxygen concentrator, cylinders or liquid oxygen and administered mainly through nasal prongs. The oxygen dose (l/min) is titrated aiming at a PaO2 on oxygen > 8 kPa in accordance with current routine practice and management guidelines.
  Interventions: Drug: LTOT 24 h/day
- LTOT 15 h/day (control) (Active Comparator): Long-term oxygen therapy (LTOT) prescribed 15 h/day. The LTOT is provided according to standard clinical practice using oxygen concentrator, cylinders or liquid oxygen and administered mainly through nasal prongs. The oxygen dose (l/min) is titrated aiming at a PaO2 on oxygen > 8 kPa in accordance with current routine practice and management guidelines.
  Interventions: Drug: LTOT 15h/day

INTERVENTIONS:
Drug: LTOT 24 h/day — LTOT prescribed for 24 h/day.
  Other Names: Long-term oxygen therapy prescribed continuously (24 h/day)
  Arms: LTOT 24 h/day (intervention)
Drug: LTOT 15h/day — : LTOT prescribed for 15 h/day. The patient is instructed to use LTOT during sleep and not to use LTOT for about 9 hours during daytime, totalling 15 h/day.
  Other Names: Long-term oxygen therapy prescribed for 15 h/day
  Arms: LTOT 15 h/day (control)

SUMMARY:
Multicenter, phase IV, non-superiority, registry-based, randomized controlled trial. Patients starting long-term oxygen therapy (LTOT) are randomized between LTOT prescribed 24 h/day or 15 h/day using the Swedish Register for Respiratory Failure (Swedevox). Clinical follow-up and concurrent treatments are according to routine clinical practice. The main endpoints of mortality, hospitalizations, and incident disease are assessed using Swedish registry data, with expected complete follow-up. Patient-reported outcomes are assessed using a posted questionnaire at 3 and 12 months. The study is managed by the Uppsala Clinical Research Centre (UCR).

DETAILED DESCRIPTION:
BACKGROUND:

LTOT given 15 h/day or more improves the survival time in patients with chronic daytime hypoxemia due to chronic obstructive pulmonary disease (COPD) based on two randomized trials; the 'Continuous or Nocturnal Oxygen Therapy' Trial (NOTT) published in 1980 [1] and the Medical Research Council (MRC) trial published in 1981.[2] International guidelines recommend that LTOT is prescribed continuously (24 h/day), which is based on an observational, unadjusted comparison of the treatment arms of the MRC and NOTT studies only. [3] However, LTOT 24 h/day may place an unnecessary burden on patients in terms of increased dependence, isolation, side effects and restricted activity.[3, 4] Data from the National Swedish Registry for Respiratory Failure (Swedevox) indicate no survival benefit from LTOT 24 vs 15 h/day (Figure 1). No randomized trial has evaluated the additional benefit of longer daily duration of LTOT above 15 h/day.[4] Studies on the effect of LTOT are also lacking for diseases other than COPD, such as pulmonary fibrosis, yet LTOT is given in these conditions according to the same criteria as in COPD in clinical practice.[4]

IMPORTANCE:

This will be the first R-RCT in respiratory medicine and the largest trial of LTOT to date. If LTOT 24 h/day is found to be superior to 15 h/day, this will confirm the importance of oxygen therapy in chronic respiratory failure and the importance of implementing services to optimize the daily duration of LTOT. If LTOT 24 h/day is non-superior to 15 h/day, this supports that patients safely can be free of supplemental oxygen for up to nine hours per day. This trial will also be the first to evaluate effects of LTOT on symptoms and HRQOL, effects in patients with moderate hypoxemia and in diseases other than COPD. This study will have direct impact on research and clinical management.

AIM:

Long-term oxygen therapy (LTOT) 24 h/day is recommended to prolong survival time in severe hypoxemia but may be burdensome and evidence of its additional benefit compared with LTOT 15 h/day is lacking. The purpose is to determine whether LTOT prescribed continuously 24 h/day fails to reduce the rate of all-cause hospitalization or death at 1 year compared with LTOT 15 h/day. The aim is improved evidence-based treatment in chronic hypoxemia.

OBJECTIVES:

Primary: To determine whether oxygen prescribed 24 h/day compared with 15 h/day in patients starting LTOT fails to improve rate of all-cause mortality or death at 1 year. Secondary objectives: evaluate between-group differences in overall and cause-specific mortality (respiratory and cardiovascular deaths); overall and cause-specific hospitalization rate; incident cardiovascular disease; breathlessness; fatigue; self-reported physical activity; health-related quality of life; cognition; measured oxygen adherence; and patient preference to continue treatment.

ANALYSIS:

Primary analysis: In all randomized patients according to the intention-to-treat and per protocol principles. Secondary analyses: In patients with severe resting hypoxemia (PaO2 < 7.4 kPa breathing air); moderate resting hypoxemia (PaO2 7.4 to 8.0 kPa breathing air); COPD verified by spirometry (FEV1/FVC < 0.7 after bronchodilation); and in patients with other conditions than COPD.

STUDY DESIGN:

Multicenter, single-blinded (analyst), effectiveness, phase IV, register-based, randomized controlled trial (R-RCT). Patients starting LTOT are randomized between oxygen prescribed 24 h/day or 15 h/day using the Swedevox registry. Clinical follow-up and concurrent treatments are according to routine clinical practice. The main endpoints of mortality, hospitalizations, and incident disease are assessed using Swedish registry data, with expected complete follow-up. Patient-reported outcomes are assessed using a postal questionnaire at 3 months. The study is managed by the Uppsala Clinical Research Centre (UCR)

Investigational products, dosage and mode of administration: Patients are randomized between two daily durations of oxygen used in current clinical practice: LTOT 24 h/day (intervention) or 15 h/day (control). The LTOT is provided according to standard clinical practice using oxygen concentrator, cylinders or liquid oxygen and administered mainly through nasal prongs. The oxygen dose (l/min) is titrated aiming at a PaO2 on oxygen > 8 kPa in accordance with current routine practice and management guidelines.

Duration of treatment: Throughout LTOT. Primary endpoint is at 1 year after randomization.

STATISTICAL METHODS:

Statistical methods: The primary analysis is according to the intention to treat (ITT) principle and the per protocol (PP) principle. Secondary analyses are according to the PP principle. The primary endpoint of the composite event of death or 1st hospitalization is analyzed with Cox´s proportional hazards model. Hospitalizations are analyzed using Fine Gray regression accounting for death as competing event. Other secondary endpoints are analyzed using two-sided Student's t-tests for continuous variables (including HRQOL, breathlessness, cognition, fatigue, activity, and health care usage) and chi-2 test for categorical variables (causes of death, cognition, treatment preference). Correlational analyses, including of factors predictive of the primary and secondary outcomes will be conducted using linear regression (continuous outcomes), logistic regression (categorical outcomes), and Cox and Fine-Gray regression models (time to event outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Severe resting hypoxemia (PaO2 < 7.4 kPa or oxygen saturation < 88% breathing air), or PaO2 < 8.0 kPa on air and either signs of heart failure or polycythemia (EVF > 0.54).

Exclusion Criteria:

* Smoking or contact with open fire
* Other inability to safely comply with LTOT
* Already on LTOT for more than 28 days
* Inability to comply with any of the study interventions as judged by the responsible oxygen staff
* Opt out from being registered in Swedevox
* Inability to give informed written consent to participate in the study as judged by the oxygen responsible staff
* Lack of Swedish identification number
* Previous participation in the study.

Patient populations that will be evaluated:

* Primary analysis: In all randomized patients according to the intention-to-treat and per protocol principles.
* Secondary analyses: In patients with 1) PaO2 (air) < 7.4 kPa; 2) PaO2 (air) 7.4 to 8.0 kPa; 3) COPD verified by spirometry (COPD as primary diagnosis and FEV1/FVC < 0.7 after bronchodilation); 4) and in patients with a primary diagnosis other than COPD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
All-cause hospitalization or mortality rate | 1 year
  To determine whether oxygen prescribed 24 h/day compared with 15 h/day in patients with chronic obstructive pulmonary disease (COPD) and severe hypoxemia improves the rate of all-cause hospitalization or mortality at 1 year.

SECONDARY OUTCOMES:
All-cause mortality rate | 3 months and 12 months
  Between-group difference in deaths from all causes
Mortality rate from respiratory disease | 3 months and 12 months
  Between-group difference in deaths from respiratory disease
Mortality rate from cardiovascular disease | 3 months and 12 months
  Between-group difference in deaths from cardiovascular disease
Hospitalization rate from all causes | 3 months and 12 months
  Between-group difference in hospitalization rate from all causes
Hospitalization rate with a primary diagnosis of respiratory disease | 3 months and 12 months
  Between-group difference in hospitalization rate with a primary diagnosis of respiratory disease
Hospitalization rate with a primary diagnosis of cardiovascular disease | 3 months and 12 months
  Between-group difference in hospitalization rate with a primary diagnosis of cardiovascular disease
Rate of an incident diagnosis of cardiovascular disease | 3 months and 12 months
  Between-group difference in rate of an incident diagnosis of cardiovascular disease
Self-reported questionnaire data on oxygen use | 3 months and 12 months
  Between-group difference in data from postal questionnaire on self-reported oxygen utilization (group percentages)
Self-reported questionnaire data on physical activity | 3 months and 12 months
  Between-group difference in data from postal questionnaire on self-reported physical activity (group percentages)
Self-reported questionnaire data on LTOT continuation | 3 months and 12 months
  Between-group difference in data from postal questionnaire on preference of continuing the LTOT (group percentages)
Self-reported questionnaire data on breathlessness (MDP scale) | 3 months and 12 months
  Between-group difference in data from postal questionnaire on breathlessness; Multidimensional Dyspnea Profile (MDP) scale. One item (A1) assesses the unpleasantness of dyspnoea on a 0-10 visual numerical scale anchored by "neutral" (0) and "unbearable" (10). Five items assess the sensory dimension of dyspnoea, both in terms of quality and intensity (on a scale of 0-10). Five items assess the affective dimension of dyspnoea, also in terms of quality and intensity (on a scale of 0-10).
  Two domain scores are calculated: an "immediate perception domain" score (S) as the sum of A1 intensity and the intensities of the five sensory descriptors; and an "emotional response domain" score (A2) as the sum of the five emotional descriptors. The median (IQR) ratings will be compared betwwen the groups.
Self-reported questionnaire data on breathlessness (mMRC scale) | 3 months and 12 months
  Between-group difference in data from postal questionnaire on breathlessness; modified Medical Research Council (mMRC) scale. measure the degree of disability that breathlessness poses on day-to-day activities on a scale from 0 to 4: 0, no breathlessness and 5 worse breathlessness. Percentages and mean scores are reported.
Self-reported questionnaire data on fatigue (FACIT-Fatigue) | 3 months and 12 months
  Between-group difference in data from postal questionnaire on fatigue; Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue scale is a 13 item questionnaire measured on a 4-point Likert scale (0 = not at all; 4 = very much). All items are summed to create a single fatigue total score with a range from 0 to 52, where higher scores indicate better functioning or less fatigue.
Self-reported questionnaire data on cognition (BAS) | 3 months and 12 months
  Between-group difference in data from postal questionnaire on cognition self-report; Informant Questionnaire on Cognitive Decline in the Elderly (IQCODE-SR) consists of 16-items (score range, 1.0-5.0; where 1=much better and 5=much worse). Total score is used.
Self-reported questionnaire data on HRQOL (CAT) | 3 months and 12 months
  Between-group difference in data from postal questionnaire on HRQOL; COPD Assessment test (CAT) consists of 8 items; 0-5 scale with higher scores indicating worse outcome and total scores ranging between 0 and 40. Mean scores are reported.
Self-reported questionnaire data on HRQOL (EQ-5D-5L) | 3 months and 12 months
  Between-group difference in data from postal questionnaire on HRQOL; EuroQol five-dimensional descriptive system (EQ-5D-5L) describing health on the dimensions of mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Scores are graded into 'no problems', 'slight problems', 'moderate problems', 'severe problems' and 'extreme problems/unable to. Mean scores are reported.
Self-reported questionnaire data on treatment response (GIC) | 3 months and 12 months
  Between-group difference in data from postal questionnaire; Global impression of change (GIC) is a 7-point descriptive scale: ranging from 1 to 7 with 1 being very much improved and 7 very much worse. Mean scores are reported.
Health care utilization | 3 months and 12 months
  Between-group difference in number of hospitalizations; number of outpatient visits and Emergency Department visits and Other medication use and cost through national registries (National Inpatient Register; National Outpatient Care Register; National Patient Register; Prescribed Drug Register)

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Ekström, MD, PhD, Principal Investigator — Blekinge County Council Hospital
Locations (2):
- Sweden (2):
  - Blekinge hospital, Karlskrona, Blekinge County
  - Örebro University Hospital, Örebro

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Continuous or nocturnal oxygen therapy in hypoxemic chronic obstructive lung disease: a clinical trial. Nocturnal Oxygen Therapy Trial Group. Ann Intern Med. 1980 Sep;93(3):391-8. doi: 10.7326/0003-4819-93-3-391. PMID 6776858
- [Background] Long term domiciliary oxygen therapy in chronic hypoxic cor pulmonale complicating chronic bronchitis and emphysema. Report of the Medical Research Council Working Party. Lancet. 1981 Mar 28;1(8222):681-6. PMID 6110912
- [Background] Anthonisen NR. Prognosis in chronic obstructive pulmonary disease: results from multicenter clinical trials. Am Rev Respir Dis. 1989 Sep;140(3 Pt 2):S95-9. doi: 10.1164/ajrccm/140.3_Pt_2.S95. No abstract available. PMID 2675713
- [Background] Hardinge M, Annandale J, Bourne S, Cooper B, Evans A, Freeman D, Green A, Hippolyte S, Knowles V, MacNee W, McDonnell L, Pye K, Suntharalingam J, Vora V, Wilkinson T; British Thoracic Society Home Oxygen Guideline Development Group; British Thoracic Society Standards of Care Committee. British Thoracic Society guidelines for home oxygen use in adults. Thorax. 2015 Jun;70 Suppl 1:i1-43. doi: 10.1136/thoraxjnl-2015-206865. PMID 25870317
- [Derived] Ekstrom M, Andersson A, Papadopoulos S, Kipper T, Pedersen B, Kricka O, Sobrino P, Runold M, Palm A, Blomberg A, Hamed R, Lindberg E, Sundberg B, Hadziosmanovic N, Bjorklund F, Janson C, McDonald CF, Currow DC, Sundh J; REDOX Collaborative Research Group. Long-Term Oxygen Therapy for 24 or 15 Hours per Day in Severe Hypoxemia. N Engl J Med. 2024 Sep 19;391(11):977-988. doi: 10.1056/NEJMoa2402638. Epub 2024 Sep 10. PMID 39254466
- [Derived] Sundh J, Bornefalk-Hermansson A, Ahmadi Z, Blomberg A, Janson C, Currow DC, McDonald CF, McCaffrey N, Ekstrom M. REgistry-based randomized controlled trial of treatment and Duration and mortality in long-term OXygen therapy (REDOX) study protocol. BMC Pulm Med. 2019 Feb 26;19(1):50. doi: 10.1186/s12890-019-0809-7. PMID 30808321
- See also: Swedish National Register for Respiratory Failure (Swedevox). Annual report. 2014. [Accessed 19 February 2016] — http://www.ucr.uu.se/swedevox/

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-05-10): https://cdn.clinicaltrials.gov/large-docs/04/NCT03441204/SAP_000.pdf